CLINICAL TRIAL: NCT04607616
Title: Interactive Guidance Therapy With Video Feed-back of Parent and Child With Autism Spectrum Disorder
Acronym: GIETSA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ville Evrard Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: APHP180671; 2019-A02707-50 (Other: ID-RCB)
Record Dates: First submitted 2020-07-01; First posted 2020-10-29 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Autism Spectrum Disorders
Keywords: Autism Spectrum Disorders; Interactive guidance therapy; Video feed-back
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Growth and Development

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 3 baselines sessions Treatment As Usual (TAU) (Experimental): Patients received 3 baseline sessions before interactive guidance therapy
  Interventions: Behavioral: Baseline sessions TAU; Behavioral: Interactive guidance therapy; Diagnostic Test: Developmental and diagnostic assessments; Behavioral: Developmental assessment -Parental scales; Behavioral: Qualitative analysis
- 4 baselines sessions TAU (Experimental): Patients received 4 baseline sessions before interactive guidance therapy
  Interventions: Behavioral: Baseline sessions TAU; Behavioral: Interactive guidance therapy; Diagnostic Test: Developmental and diagnostic assessments; Behavioral: Developmental assessment -Parental scales; Behavioral: Qualitative analysis
- 5 baselines sessions TAU (Experimental): Patients received 5 baseline sessions before interactive guidance therapy
  Interventions: Behavioral: Baseline sessions TAU; Behavioral: Interactive guidance therapy; Diagnostic Test: Developmental and diagnostic assessments; Behavioral: Developmental assessment -Parental scales; Behavioral: Qualitative analysis
- 6 baselines sessions TAU (Experimental): Patients received 6 baseline sessions before interactive guidance therapy
  Interventions: Behavioral: Baseline sessions TAU; Behavioral: Interactive guidance therapy; Diagnostic Test: Developmental and diagnostic assessments; Behavioral: Developmental assessment -Parental scales; Behavioral: Qualitative analysis
- 7 baselines sessions TAU (Experimental): Patients received 7 baseline sessions before interactive guidance therapy
  Interventions: Behavioral: Baseline sessions TAU; Behavioral: Interactive guidance therapy; Diagnostic Test: Developmental and diagnostic assessments; Behavioral: Developmental assessment -Parental scales; Behavioral: Qualitative analysis
- 8 baselines sessions TAU (Experimental): Patients received 8 baseline sessions before interactive guidance therapy
  Interventions: Behavioral: Baseline sessions TAU; Behavioral: Interactive guidance therapy; Diagnostic Test: Developmental and diagnostic assessments; Behavioral: Developmental assessment -Parental scales; Behavioral: Qualitative analysis

INTERVENTIONS:
Behavioral: Baseline sessions TAU — TAU consists of sessions lasting around one/one and a half hour ; the consultant is practicing as usual. The interventions focus on child's behavior, parent infant relationship, with moments of play with the child, advices, informations about child development and Autism.
Behavioral: Interactive guidance therapy — The objective is to reinforce the identification, deciphering, interpretation, and answer to child's signals by the parent, in order to to promote a synchronous and attuned response to the child's needs.
  Sessions last around one/one and a half hour. Parent plays 7-10 minutes with the child, in the presence of the therapist, with toys chosen according to the child's developmental stage. Then therapist proposes an immediate viewing of the play session. The therapist selects short moments of positive interaction. He has determined a " focus ", depending on the play, previous sessions, the child's difficulties and parent's interventions. He accompanies, guides and supports the parent to describe the interaction, the alternance in play, joint attention, shared affect, in a co-construction: the parent discovers the child's and his own skills.
Diagnostic Test: Developmental and diagnostic assessments — MSEL, CARS, ECAR, CIM10, DMS5, ADOS, ADIR
Behavioral: Developmental assessment -Parental scales — Vineland II, IFDC, IDE
Behavioral: Qualitative analysis — Interpretative Phenomenological Analysis. Parents' semi structured interview about the Interactive Guidance experience. Qualitative analysis of transcripts (recurrent themes, meta themes).

SUMMARY:
The purpose of this study is to assess the effect of Interactive Guidance Therapy with video feed back (IGT) of parent and child with Autism Spectrum Disorder, under three years of age, using a Single Case Experimental Design (SCED) with multiple baseline across subjects, multicentric, randomized, with multiple replications, blinded scored

DETAILED DESCRIPTION:
The purpose of this study is to assess the effect of Interactive Guidance Therapy with video feed back (IGT) of parent and child with Autism Spectrum Disorder, under three years of age, using a Single Case Experimental Design.

Early Interventions in Autism Spectrum Disorders (ASD) undergo a major development. The investigators identify three generations of early support: 1) Behavioral studies ; 2) Early Intensive Behavioral Interventions (EIBI), inspired by ABA, focused on targeted ASD disorders 3) Naturalistic Behavioral Developmental Behavioral Interventions (NDBI), more ecological, focused on the child's skills.

Among them, methods of video feedback target parental sensitivity (identification, interpretation, response, contingency and synchrony). The VIPP (Video Interactive Positive Parenting) in children less than one year of age, has shown moderate and long term effects on parent-child interaction. The PACT (Preschool Autism Communication Trial) showed immediate and in the long term effects on the synchronization of the parental response, the child initiation, less importantly on the joint attention, and on the autistic symptoms. The dyadic communication allows for changes in autistic symptoms.

Interactive guidance is a brief video-feedback therapy, based on the analysis of "the here and now" with the parent (s), of videotaped interactions with their child. The objective is to strengthen parental skills, their sensitivity, their ability to decipher and respond to the specific needs of their child.

The interest of IGT in the field of ASD, compared to VIPP and PACT, is to offer a standardized feedback intervention adapted to each dyad, according to the child's and parents skills and difficulties, structured on the "here and now" more than on a predetermined sequence of goals.

The investigators use the Single Case Experimental Design (SCED) with multiple baseline across subjects, multicentric, randomized, with multiple replications, blinded scored.

They expect

* to improve the interactive and communicative basic skills of the child, soon after the ASD diagnosis, by accompanying the parents in the identification and understanding of their child's disorders.
* to propose a method highlighting parental skills, in a collaborative and pleasant way
* To increase the parental alliance in the implementation of a tailored intervention for the child
* To facilitate access to healthcare and reduce the parental wandering in the implementation of intervention

ELIGIBILITY:
Inclusion Criteria:

* 18 months to 3 years child at screening
* Child with a diagnosis of Autism Spectrum Disorder (DSM 5) or pervasive Developmental Disorder (ICD 10)
* Child with ADI R and ADOS-2 fulfilling the criteria for TSA / PDD at diagnosis
* Developmental age > 12 months in motility with the Brunet-Lézine test
* Child with availability of parent most present in daily life, only this parent participating directly in play sessions
* Signed Informed consent form by both parents
* Patient affiliated to the health insurance system

Exclusion Criteria:

* Level of language in French of parents insufficient to benefit from the care and fill in the questionnaires
* Psychiatric parental pathology interfering with interactions with the child, qualitatively assessed by the referring psychiatrist
* Severe sensory illness of the child (blindness, deafness, degenerative disease)

Ages: 18 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2021-03-26 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of time spent in a joint attention situation | Up to 15 months
  Coordinated Joint Attention (COJ) rate is evaluated during the parents-child play-time
Percentage of time spent in a joint attention situation | Up to 15 months
  Supported Joint Attention (SUJ) rate is evaluated during the parents-child play-time

SECONDARY OUTCOMES:
Parent-child interactive features/ joint attention | Up to 15 months
  - SUJ and COJ rate initiated by child
Parent-child interactive features / DCMA scale | Up to 15 months
  - DCMA: dyadic communication measure in autism
Parent-child interactive features / Parental synchrony | Up to 15 months
  - number of parental responses in synchrony with child
Parent-child interactive features / Communication | Up to 15 months
  - Number conversational turns of speech between the child and the parent
Parent-child interactive features / Initiation of communication | Up to 15 months
  - Initiation of communication by the child with the parent : in proportion to the child's acts of communication
Child development / MSEL | Up to 15 months
  - MSEL : is Mullen Scale of Early Learning evaluated at inclusion visit, guidance session 1, guidance session 10 and guidance session 15
Child development / CDI | Up to 15 months
  - CDI is Child Development Inventory evaluated at inclusion visit, guidance session 1, guidance session 10 and guidance session 15
Child development / IFDC | Up to 15 months
  - IFDC is French adaptation of MacArthur-Bates Communicative Development Inventories evaluated at inclusion visit, guidance session 1, guidance session 10 and guidance session 15
Autistic Symptoms / CARS | Up to 15 months
  CARS is Childhood Autism Rating Scale evaluated at inclusion visit, guidance session 1, guidance session 10 and guidance session 15
Autistic Symptoms ECAR | Up to 15 months
  ECA R is "Evaluation des comportements autistiques Révisée" Scale evaluated at inclusion visit, guidance session 1, guidance session 10 and guidance session 15
Autistic Symptoms ADOS-2 | Up to 15 months
  ADOS-2 is Autism diagnostic observation Schedule evaluated at inclusion visit, guidance session 1, guidance session 10 and guidance session 15
Autistic Symptoms ADIR | Up to 15 months
  ADI R is Autism Diagnosis Interview Revised evaluated at inclusion visit, guidance session 1, guidance session 10 and guidance session 15
Adaptive behavior of the child | Up to 15 months
  Vineland 2 Scale evaluated at inclusion visit, guidance session 1, guidance session 10 and guidance session 15
Change process | Up to 15 months
  Psychotherapy Process Q-set evaluated at baseline visit 1 and last baseline visit (depend of randomization), guidance session 1 and guidance session 10
Content analysis of guidance session by parent | At 16 months
  Targeted interview of parents with the psychologist on the content of guidance session

CONTACTS AND LOCATIONS:
Overall Officials: Benoit QUIROT, MD, Study Director — EPS Ville Evrard
Locations (4):
- France (4):
  - Hôpital Saint Eloi, Montpellier
  - Hôpital Ville Evrard, Montreuil
  - Hôpital Pitié Salpétriere, Paris
  - Hôpital Necker Enfants Malades, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. McDonough S. Interaction guidance. Treat Parent-infant Relatsh Probl Strateg Interv. 2004;79-96.
- [Background] 2. McDonough SC. Promoting positive early parent-infant relationships through interaction guidance. Child Adolesc Psychiatr Clin N Am. 1995;4(3):661-72.
- [Background] Rusconi-Serpa S, Sancho Rossignol A, McDonough SC. Video feedback in parent-infant treatments. Child Adolesc Psychiatr Clin N Am. 2009 Jul;18(3):735-51. doi: 10.1016/j.chc.2009.02.009. PMID 19486848